CLINICAL TRIAL: NCT03177395
Title: A Randomised Open Label Exploratory, Safety and Tolerability Study With PP100-01 in Patients Treated With the 12-hour Regimen of N-Acetylcysteine for Paracetamol/Acetaminophen Overdose (The POP Trial)
Brief Title: PP100-01 (Calmangafodipir) for Overdose of Paracetamol
Acronym: POP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egetis Therapeutics (Industry)
Collaborators: University of Edinburgh (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP100-001
Record Dates: First submitted 2017-05-23; First posted 2017-06-06 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Paracetamol Overdose
MeSH Terms: interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetylcysteine (N-acetylcysteine; NAC) (No Intervention): NAC infusion 100mg/kg in 200ml 'loading dose' at timepoint '0'. 12 hour NAC regime will be continued with the second dose: 200mg/kg NAC in 1000ml i.v. over 10hr as per standard care protocol in NHS Lothian.
- PP100-01 (Calmangafodipir)+ NAC (Experimental): In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  * Group A: PP100-01 (2 umol/kg calmangafodipir) after the "loading" dose of NAC
  * Group B: PP100-01 (5 umol/kg calmangafodipir) after the "loading" dose of NAC
  * Group C: PP100-01 (10 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  Interventions: Drug: PP100-01 (calmangafodipir); Drug: Acetylcysteine

INTERVENTIONS:
Drug: PP100-01 (calmangafodipir) — PP100-01
  Other Names: PP100-01
  Arms: PP100-01 (Calmangafodipir)+ NAC
Drug: Acetylcysteine — NAC
  Other Names: N-acetylcysteine
  Arms: PP100-01 (Calmangafodipir)+ NAC

SUMMARY:
Investigate the safety and tolerability of PP100-01 add-on treatment to the 12hr NAC treatment regime in patients treated for paracetamol/acetaminophen overdose (POD) when NAC treatment is initiated before 24hours post POD.

DETAILED DESCRIPTION:
The study will be an open label, randomised, exploratory, rising dose design, NAC controlled, phase 1 safety and tolerability study in patients treated with NAC for paracetamol/acetaminophen overdose.

Entry into the study will depend on the patient's blood results confirming the need for NAC. A total of 24 patients will be assigned into one of 3 dosing cohorts of 8 patients (N=6 for PP100-01 and NAC; N=2 for NAC alone).

The study will primarily evaluate safety and tolerability for treatment with PP100-01 in combination with NAC as compared to NAC alone.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with capacity admitted to hospital within 24 hrs either a single acute POD or more than one dose of paracetamol (staggered) and deemed to require treatment with NAC.
2. Provision of written informed consent
3. Males and females of at least 16 years of age

Exclusion Criteria:

1. Patients that do not have the capacity to consent to participate in the study
2. Patients detained under the Mental Health Act or deemed unfit by the Investigator to participate due to mental health.
3. Patients with known permanent cognitive impairment
4. Patients who are pregnant or nursing
5. Patients who have previously participated in the study
6. Unreliable history of POD
7. Patients presenting after 24hrs of POD
8. Patients who take anticoagulants (e.g. warfarin) therapeutically or have taken an overdose of anticoagulants
9. Patients who, in the opinion of the responsible clinician/nurse, are unlikely to complete the full course of NAC e.g. expressing wish to self-discharge
10. Prisoners
11. Non-English speaking patients. (Study information material will only be produced in English in view of the known and stable demographic of the Edinburgh self-harm population).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Dear, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, City Of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrison EE, Oatey K, Gallagher B, Grahamslaw J, O'Brien R, Black P, Oosthuyzen W, Lee RJ, Weir CJ, Henriksen D, Dear JW; POP Trial Investigators. Principal results of a randomised open label exploratory, safety and tolerability study with calmangafodipir in patients treated with a 12 h regimen of N-acetylcysteine for paracetamol overdose (POP trial). EBioMedicine. 2019 Aug;46:423-430. doi: 10.1016/j.ebiom.2019.07.013. Epub 2019 Jul 13. PMID 31311721
- [Derived] POP Trial Investigators; Dear J. Randomised open label exploratory, safety and tolerability study with calmangafodipir in patients treated with the 12-h regimen of N-acetylcysteine for paracetamol overdose-the PP100-01 for Overdose of Paracetamol (POP) trial: study protocol for a randomised controlled trial. Trials. 2019 Jan 8;20(1):27. doi: 10.1186/s13063-018-3134-1. PMID 30621764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Studied period: 05 June 2017 to 08 August 2018 Study centres: Edinburgh Clinical Trials Unit (ECTU) The Emergency Medicine Research Group Edinburgh (EMERGE)
Pre-assignment Details: Adults within 24 h of a paracetamol overdose that required NAC. Within each of 3 sequential cohorts, participants were randomly assigned, with concealed allocation, to NAC and a single intravenous calmangafodipir dose (n=6/dose) or NAC alone (n=2). Calmangafodipir doses were 2, 5, or 10 μmol/kg. Participants, study and clinical teams not blinded
Groups:
- Group A: PP100-01 (Calmangafodipir 2 μmol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (2 μmol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
- Group B: PP100-01 (Calmangafodipir 5 μmol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (5 μmol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
- Group C: PP100-01 (Calmangafodipir 10 μmol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (10 μmol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
Period: Overall Study
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 μmol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 μmol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 μmol/kg)+ NAC
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 24 participants randomised to the study. All participants received the full dose of PP100-01 according to the allocated dosing cohort where randomised to PP100-01 treatment and all participants received as a minimum 12 hours of NAC treatment (loading dose, plus further 10 hours). Total dose was adjusted according to participant weight
Groups:
- Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (2 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
- Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (5 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
- Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  • Group B: PP100-01 (5 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 (10 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
- Total: Total of all reporting groups
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 6 | 6 | 23
  >=65 years | 0 | 1 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (12.5) | 42.5 (13.1) | 42.7 (12.7) | 22.7 (3.3) | 35.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 3 | 13
  Male | 4 | 2 | 2 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 6 | 6 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 24
Time from ingestion of paracetamol to hospital presentation [Mean (Standard Deviation); unit: hours] | 8.8 (6.2) | 6.0 (6.2) | 5.8 (7.2) | 4.9 (5.2) | 6.4 (6.2)
Type of overdose [Count of Participants; unit: Participants]
  Acute, ≤8 h to NAC | 2 | 4 | 4 | 4 | 14
  Acute, >8 h to NAC | 3 | 2 | 2 | 1 | 8
  Staggered intentional | 0 | 0 | 0 | 1 | 1
  Supra-therapeutic | 1 | 0 | 0 | 0 | 1
Presentation paracetamol concentration [Mean (Standard Deviation); unit: mg/L] | 76 (81) | 127 (90) | 74 (44) | 127 (47) | 101 (66)
Total paracetamol ingested [Mean (Standard Deviation); unit: mg/kg] | 185 (156) | 235 (77) | 229 (72) | 397 (476) | 262 (195)
Time from ingestion of paracetamol to start of NAC treatment [Mean (Standard Deviation); unit: hours] | 12.1 (5.2) | 9.8 (6.5) | 10.2 (6.9) | 8.6 (4.1) | 10.2 (5.7)
Time from ingestion of paracetamol to start of calmangafodipir [Mean (Standard Deviation); unit: hours] | NA (NA) — No IMP given | 12.6 (6.8) | 10.8 (4.1) | 11.8 (5.4) | 11.7 (5.4)
Any other drug ingested [Count of Participants; unit: Participants]
  Yes | 5 | 4 | 5 | 5 | 19
  No | 1 | 2 | 1 | 1 | 5
Serum creatinine [Mean (Standard Deviation); unit: μmol/L] | 74.7 (11.0) | 67.5 (13.3) | 67.3 (17.2) | 69.5 (13.1) | 69.8 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Safety Events
Description: Adverse Events and Serious Adverse Events
Time Frame: 90 days
Population: In addition to paracetamol overdose, 19 out of the 24 randomised participants reported taking overdoses of other medicines in addition to the paracetamol. All treatment groups included participants with paracetamol only overdoses and mixed overdoses
Measure: Number; unit: participants
Groups:
- Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  * Group A: PP100-01 (2 umol/kg calmangafodipir) after the "loading" dose of NAC PP100-01 (5 umol/kg calmangafodipir) after the "loading" dose of NAC
  * Group C: PP100-01 (10 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
- Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (10 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Any Adverse event | 6 | 6 | 6 | 6
  Any serious adverse event | 2 | 4 | 2 | 3
  Adverse event after commencement of NAC treatment | 6 | 5 | 6 | 6
  Serious AE after commencement of NAC treatment | 1 | 1 | 1 | 2
  Adverse event where outcome was death | 0 | 0 | 1 | 0
  Adverse event unrelated to NAC | 3 | 5 | 3 | 5
  Adverse event possibly related to NAC | 2 | 2 | 2 | 2
  Adverse event probably related to NAC | 3 | 2 | 3 | 2
  Adverse event definitely related to NAC | 2 | 3 | 1 | 1
  Adverse event unrelated to PP100-01 | 6 | 6 | 5 | 6
  Adverse event possibly related to PP100-01 | 0 | 4 | 2 | 2
  Adverse event probably related to PP100-01 | 0 | 0 | 0 | 0
  Adverse event definitely related to PP100-01 | 0 | 0 | 0 | 0
  Any suspected unexpected serious adverse reaction | 0 | 0 | 0 | 1
  SUSAR to NAC | 0 | 0 | 0 | 0
  SUSAR to PP100-01 | 0 | 0 | 0 | 1
  SUSAR to NAC and PP100-01 | 0 | 0 | 0 | 0

2. Secondary Outcome: ALT(U/L)
Description: The alanine aminotransferase (ALT) test is a blood test that checks for liver damage.
Time Frame: Baseline
Measure: Geometric Mean (Standard Deviation); unit: U/L
Groups:
- Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC: In addition to the standard care NAC regime, participants will be allocated into a dosing cohort to receive:
  PP100-01 (5 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 (10 umol/kg calmangafodipir) after the "loading" dose of NAC
  PP100-01 treatment is administered intravenously over 5 minutes.
  PP100-01 (calmangafodipir): PP100-01
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 42.5 (3.6) | 24.6 (2.1) | 29.4 (2.3) | 17.7 (1.5)

3. Secondary Outcome: ALT(U/L)
Description: The alanine aminotransferase (ALT) test is a blood test that checks for liver damage.
Time Frame: 10 hours
Population: All 24 participants received the full dose of PP100-01 according to the allocated dosing cohort, all participants received as a minimum 12 hours of NAC treatment (loading dose, plus further 10 hours). For both PP100-01 and NAC total dose was adjusted according to participant weight
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 41.4 (3.3) | 22.9 (1.8) | 25.3 (2.1) | 15.0 (1.3)

4. Secondary Outcome: ALT(U/L)
Description: The alanine aminotransferase (ALT) test is a blood test that checks for liver damage.
Time Frame: 20 hours
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 43.3 (3.8) | 20.4 (1.9) | 25.4 (1.8) | 16.4 (1.5)

5. Secondary Outcome: INR
Description: international normalised ratio (INR) characterise acute liver injury (ALI) and failure (ALF)
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 5 | 6 | 6
ratio | 1.02 (0.04) | 1.00 (0.12) | 0.98 (0.04) | 1.05 (0.14)

6. Secondary Outcome: INR
Description: international normalised ratio (INR) characterise acute liver injury (ALI) and failure (ALF)
Time Frame: 10 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.30 (0.18) | 1.17 (0.20) | 1.20 (0.00) | 1.22 (0.25)

7. Secondary Outcome: INR
Description: international normalised ratio (INR) characterise acute liver injury (ALI) and failure (ALF)
Time Frame: 20 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio | 1.18 (0.21) | 1.07 (0.19) | 1.08 (0.04) | 1.22 (1.17)

8. Secondary Outcome: INR
Description: international normalised ratio (INR) characterise acute liver injury (ALI) and failure (ALF)
Time Frame: value at 20 hours divided by baseline value for each patient
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 5 | 6 | 6
ratio | 1.15 (1.17) | 1.07 (1.12) | 1.10 (1.07) | 1.10 (1.10)

9. Secondary Outcome: Additional NAC Infusion
Description: participants required additional NAC infusions after the 12-hour NAC regimen
Time Frame: Additional NAC at 12 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  None | 3 | 5 | 6 | 6
  One | 1 | 1 | 0 | 0
  Two | 2 | 0 | 0 | 0

10. Secondary Outcome: K18 (U/L)
Description: In paracetamol overdose, the full-length variant of Keratin-18 (K-18) is released by necrotic hepatocyte death.
Time Frame: Baseline (2 hours)
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 187 (2.20) | 177 (1.82) | 193 (1.56) | 128 (1.25)

11. Secondary Outcome: K18(U/L)
Description: In paracetamol overdose, the full-length variant of Keratin-18 (K-18) is released by necrotic hepatocyte death.
Time Frame: 10 hours
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 182 (1.95) | 152 (1.56) | 170 (1.42) | 111 (1.18)

12. Secondary Outcome: K18 (U/L)
Description: In paracetamol overdose, the full-length variant of Keratin-18 (K-18) is released by necrotic hepatocyte death.
Time Frame: 20 hours
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 347 (3.18) | 229 (1.94) | 172 (1.45) | 181 (1.73)

13. Secondary Outcome: K18 (U/L)
Description: In paracetamol overdose, the full-length variant of Keratin-18 (K-18) is released by necrotic hepatocyte death.
Time Frame: Ratio - value at 20 hours divided by baseline value for each patient
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 1.85 (1.47) | 1.29 (1.89) | 0.89 (1.57) | 1.41 (1.83)

14. Secondary Outcome: ccK18 (U/L)
Description: The shorter, Caspase cleaved form of K-18 is released following hepatocyte apoptosis (programmed cell death).
Time Frame: Baseline (2 hours)
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 67 (1.99) | 45 (1.33) | 84 (1.80) | 104 (2.44)

15. Secondary Outcome: ccK18 (U/L)
Description: The shorter, Caspase cleaved form of K-18 is released following hepatocyte apoptosis (programmed cell death).
Time Frame: 10 hours
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 72 (2.24) | 53 (1.25) | 56 (1.57) | 78 (2.12)

16. Secondary Outcome: ccK18 (U/L)
Description: The shorter, Caspase cleaved form of K-18 is released following hepatocyte apoptosis (programmed cell death).
Time Frame: 20 hours
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 149 (3.34) | 66 (1.34) | 85 (1.62) | 111 (2.56)

17. Secondary Outcome: ccK18 (U/L)
Description: Caspace-cleaved Keratin-18
Time Frame: Ratio - value at 20 hours divided by baseline value for each patient
Measure: Geometric Mean (Standard Deviation); unit: U/L
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
U/L | 2.22 (1.77) | 1.49 (1.55) | 1.02 (1.79) | 1.08 (2.44)

18. Secondary Outcome: miR-122 (Delta Count)
Description: MiR-122 is a biomarker specific for liver injury and fully conserved (translational) across in vitro models, in vivo models and humans. MiR-122 is an early marker for acute liver injury which predicts a rise in ALT activity following paracetamol overdose
Time Frame: Baseline (2 hours)
Measure: Mean (Standard Deviation); unit: DCt
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
DCt | 5.58 (3.36) | 5.85 (1.50) | 4.43 (3.92) | 8.73 (2.36)

19. Secondary Outcome: miR-122 (Delta Count)
Description: as for outcome 18
Time Frame: 10 hours
Measure: Mean (Standard Deviation); unit: DCt
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
DCt | 5.41 (3.86) | 6.14 (1.99) | 5.01 (3.36) | 9.00 (1.45)

20. Secondary Outcome: miR-122 (Delta Count)
Description: as for outcome 18
Time Frame: 20 hours
Measure: Mean (Standard Deviation); unit: DCt
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
DCt | 4.85 (3.97) | 7.12 (2.26) | 4.49 (2.93) | 8.44 (1.50)

21. Secondary Outcome: miR-122 (Copies/mcL)
Description: as for outcome 18
Time Frame: Baseline (2 h)
Measure: Geometric Mean (Standard Deviation); unit: copies/mcL
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
copies/mcL | 146,363 (11.7) | 116,749 (2.4) | 194,075 (13.5) | 36,051 (3.9)

22. Secondary Outcome: miR-122(Copies/mcL)
Description: as for outcome 18
Time Frame: 10 hours
Measure: Geometric Mean (Standard Deviation); unit: copies/mcL
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
copies/mcL | 206,205 (13.0) | 109,882 (3.3) | 196,732 (9.4) | 37,066 (2.2)

23. Secondary Outcome: miR-122 (Copies/mcL)
Description: as for outcome 18
Time Frame: 20 hours
Measure: Geometric Mean (Standard Deviation); unit: copies/mcL
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
copies/mcL | 216,256 (10.8) | 57,664 (3.8) | 202,271 (7.7) | 40,745 (3.2)

24. Secondary Outcome: miR-122 (Copies/mcL)
Description: as for outcome 18
Time Frame: Ratio - value at 20 hours divided by baseline value for each patient
Measure: Geometric Mean (Standard Deviation); unit: copies/mcL
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
Number analyzed (Participants) | 6 | 6 | 6 | 6
copies/mcL | 1.48 (5.71) | 0.49 (1.98) | 1.04 (8.28) | 1.13 (2.96)

ADVERSE EVENTS:
Time Frame: Adverse events / adverse reactions were assessed at baseline, 2, 2.5, 10, 20 and 22 hours as well as ad hoc and as part of follow up. Following discharge, patients were followed up using their electronic records. AE data were collected 7, 30 and 90 days after randomisation
Arm/Group | Acetylcysteine (N-acetylcysteine; NAC) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 2/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetylcysteine (N-acetylcysteine; NAC) (N=6) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC (N=6) | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC (N=6) | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC (N=6)
cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Chest tightnes
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Nausea, vomiting
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — depressive episode;, mental health crisis;mental health issue (11006)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — seizures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetylcysteine (N-acetylcysteine; NAC) (N=6) | Group A: PP100-01 (Calmangafodipir 2 Umol/kg)+ NAC (N=6) | Group B: PP100-01 (Calmangafodipir 5 Umol/kg)+ NAC (N=6) | Group C: PP100-01 (Calmangafodipir 10 Umol/kg)+ NAC (N=6)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (3) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
heart block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 4 (4) | 4 (7) | 2 (2) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaethesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ntentional product misuse (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
substance abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/95/NCT03177395/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT03177395/SAP_001.pdf